CLINICAL TRIAL: NCT02515279
Title: A Non-Interventional Trial of Pegasys/Copegus in HCV Patients for 12 Months
Brief Title: An Observational Study of Peginterferon Alfa-2a Plus Ribavirin for Hepatitis C Virus (HCV) Infection in Austria
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22273
Record Dates: First submitted 2015-07-29; First posted 2015-08-04 (Estimated); Results first posted 2016-02-10 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Participants With Hepatitis C: All participants were treated with Peginterferon alfa-2a+Ribavirin (Pegasys/Copegus) according to the summary of product characteristics and to the investigator's discretion. The daily recommended dose for Pegasys, for the treatment of chronic Hepatitis C, was 180 micrograms once weekly by subcutaneous administration. Copegus was administered orally in doses according to the physician's decision (depending on the participant's weight and genotype). All participants were observed for 12 months.
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Peginterferon alfa-2a — 180 micrograms subcutaneous weekly for 48 weeks.
  Other Names: Pegasys
Drug: Ribavirin — 1000-1600 mg day orally for 48 weeks.
  Other Names: Copegus

SUMMARY:
This noninterventional, open-label study will observe the safety and tolerability of peginterferon alfa-2a in combination with ribavirin among Austrian participants treated for HCV infection according to routine practice.

ELIGIBILITY:
Inclusion Criteria:

* Ongoing treatment with peginterferon alfa-2a and ribavirin at the discretion of the prescribing physician
* HCV infection

Exclusion Criteria:

* None specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will enroll Austrian participants receiving peginterferon alfa-2a and ribavirin for HCV infection according to routine practice.
Sampling Method: Non-Probability Sample
Enrollment: 463 (Actual)
Dates: Start 2008-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- A.Ö. Krankenhaus Der Barmherzigen Schwestern Ried; Interne Abtl., Ried-innkreis, Austria

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants With Hepatitis C
Started | 463
Completed | 359
Not Completed | 104
Not completed — Adverse Event | 7
Not completed — Lack of Efficacy | 31
Not completed — Lost to Follow-up | 9
Not completed — Withdrawal by Subject | 18
Not completed — End-of-treatment visit not attended | 17
Not completed — Other | 22

BASELINE CHARACTERISTICS:
Population: All participants who were enrolled in the study.
Arm/Group | Participants With Hepatitis C
Number analyzed (Participants) | 463
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (13.3)
Sex/Gender, Customized [Number; unit: participants]
  Female | 151
  Male | 310
  Missing | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) and Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability or incapacity; and congenital anomaly. Percentage of participants with AEs included participants affected with both SAEs and non-SAEs.
Time Frame: Up to 6 years
Population: All participants who were enrolled in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Hepatitis C
Number analyzed (Participants) | 463
percentage of participants
  AEs | 44.28
  SAEs | 3.9

2. Primary Outcome: Percentage of Participants With End of Treatment Response
Description: Clinical response to the treatment was measured by qualitative negative polymerase chain reaction (PCR). A participant was considered to have and end of treatment response if there was undetectable Hepatitis C Virus (HCV) ribonucleic acid (RNA) after completing treatment. Participants with available PCR results were reported.
Time Frame: 12 months
Population: All participants who were enrolled in the study. N (Number of participants analysed)=participants who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Hepatitis C
Number analyzed (Participants) | 446
percentage of participants
  Participants with negative PCR | 83.8
  Participants with positive PCR | 9.7

3. Primary Outcome: Percentage of Participants With Sustained Virologic Response 24 (SVR24)
Description: Clinical response to the treatment was measured by qualitative negative polymerase chain reaction (PCR). SVR24 is defined as the percentage of participants with undetectable HCV RNA 24 weeks after completing treatment.
Time Frame: 18 months
Population: All participant who were enrolled in the study. N=number of participants evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Hepatitis C
Number analyzed (Participants) | 144
percentage of participants | 26.6

ADVERSE EVENTS:
Time Frame: up to 6 years
Description: All participant who were enrolled in the study.
Arm/Group | Participants With Hepatitis C
Serious Adverse Events (participants affected / at risk) | 18/463
Other Adverse Events (participants affected / at risk) | 148/463
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Hepatitis C (N=463)
Anaemia (Blood and lymphatic system disorders) | 8
Leukopenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Influenza like illness (General disorders) | 4
Fatigue (General disorders) | 2
Headache (Nervous system disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Depression (Psychiatric disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Syncope (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Hepatitis C (N=463)
Leukopenia (Blood and lymphatic system disorders) | 64
Anaemia (Blood and lymphatic system disorders) | 59
Thrombocytopenia (Blood and lymphatic system disorders) | 40
Fatigue (General disorders) | 39
Depression (Psychiatric disorders) | 27
Pruritus (Skin and subcutaneous tissue disorders) | 26

LIMITATIONS AND CAVEATS:
The sustained viral response that had to be filled out 6 months (or later) after the end of treatment was documented poorly due to reasons such as participants that were lost to follow-up or the study closure was before the visit date for the SVR.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.